CLINICAL TRIAL: NCT00274924
Title: Response-Adapted Therapy for Aggressive Non-Hodgkin's Lymphomas Based on Early [18F] FDG-PET Scanning
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Stage II, Stage III, or Stage IV Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455012; U10CA021115 (NIH); E3404 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Carboplatin; Cyclophosphamide; carboxypeptidase M; Doxorubicin; Etoposide; Podophyllotoxin; Ifosfamide; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (PET negative) (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine
- Group II (PET positive) (Experimental): Patients receive R-ICE comprising rituximab IV on day 1, ifosfamide IV continuously over 24 hours and carboplatin IV over 30 minutes on day 2, and etoposide IV over 2 hours on days 1-3. Patients also receive filgrastim (G-CSF) subcutaneously once daily starting on day 4 and continuing until blood counts recover. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: carboplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: ifosfamide

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously or intravenous bolus.
  Other Names: G-CSF, Neupogen, recombinant-methionyl human granulocyte-colony stimulating; factor, granulocyte colony-stimulating factor, r-metHuG-CSF.
  Arms: Group II (PET positive)
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8, Chimeric anti-CD20 monoclonal antibody, Rituxan.
Drug: carboplatin — Given IV
  Other Names: CBDCA, Paraplatin, JM-8, NSC #241240.
  Arms: Group II (PET positive)
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan, Neosar, CTX, CPM.
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin, Rubex, Adriamycin RDF, Adriamycin PFS, hydroxydaunorubicin,; hydroxydaunomycin, ADR.
  Arms: Group I (PET negative)
Drug: etoposide — Given IV
  Other Names: VP-16, VePesid, epipodophyllotoxin
  Arms: Group II (PET positive)
Drug: ifosfamide — Given IV
  Other Names: Isophosphamide, Ifex , Mitoxan , Holoxan , Naxamide ' NSC # 109724.
  Arms: Group II (PET positive)
Drug: prednisone — Taken orally
  Other Names: Deltasone, Orasone, Medicorten, Panasol-S, Liquid-Pred, others.
  Arms: Group I (PET negative)
Drug: vincristine — Given IV
  Other Names: Oncovin, Vincasar PFS vincristine sulfate, VCR, leucocristine, LCR.
  Arms: Group I (PET negative)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating patients with stage II, stage III, or stage IV diffuse large B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year progression-free survival (PFS) rate after treatment with rituximab, ifosfamide, carboplatin, and etoposide (R-ICE) in patients with bulky stage II or stage III or IV diffuse large B-cell non-Hodgkin's lymphoma who remain positron emission tomography (PET)-positive after 3 courses of rituximab, cyclophosphamide, vincristine, doxorubicin hydrochloride, and prednisone.

Secondary

* Determine the proportion of mid-treatment PET-positive patients who become PET-negative after 4 courses of R-ICE.
* Determine the PFS of mid-treatment PET-negative patients treated with these regimens.
* Determine the overall survival of patients treated with these regimens.
* Determine the toxicity of these regimens in these patients.

OUTLINE:

* Rituximab and Combination Chemotherapy (R-CHOP: R= Rituximab, C= Cyclophosphamide, H= Doxorubicin Hydrochloride (Hydroxydaunomycin), O= Vincristine Sulfate (Oncovin), P= Prednisone): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients undergo fludeoxyglucose F18 positron emission tomography (PET) scanning and conventional restaging during course 3. Based on the PET results, patients are assigned to 1 of 2 treatment groups.

  * Group I (PET negative): Patients receive 2 more courses of R-CHOP as above in the absence of disease progression or unacceptable toxicity.
  * Group II (PET positive): Patients receive Rituximab 375 mg/m2 IV Day 1, Ifosfamide 5000 mg/m2 IV over 24 hours Day 2, Carboplatin AUC 5 (max: 800 mg) IV Day 2, Etoposide 100 mg/m2 IV Days 1, 2, 3 (R-ICE), Mesna 5000 mg/m2 IV over 24 hours Day 2, and Filgrastim 5 mcg/kg/day subcutaneous (SC) Day 4 until absolute neutrophil count (ANC) recovery every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 10 years from the date of study entry.

ACCRUAL: A total of 100 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diffuse large B-cell non-Hodgkin's lymphoma

  * Bulky stage II (bulk defined as any lesion ≥ 10 cm) or stage III or IV disease
  * The following lymphoma types are excluded:

    * Primary central nervous system lymphoma
    * Transformed low-grade lymphoma (prior history of low-grade lymphoma or clear presence of low-grade lymphoma on histologic sections)
    * Primary mediastinal B-cell lymphoma or testicular lymphoma (consolidative radiotherapy is usually indicated)
    * Immunodeficiency-related lymphoma (i.e., after organ or bone marrow transplant)
* Measurable disease

  * Patient must have at least one objective measurable disease site (i.e., measurable in at least 2 perpendicular parameters)
  * Measurable disease in the liver is required if the liver is the only site of lymphoma involvement
  * Abnormal positron emission tomography scans will not constitute evaluable disease, unless verified by CT scan or other appropriate imaging
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* For patients > 50 years of age, a normal ejection fraction by ECHO or Multigated Acquisition Scan (MUGA) is required within 6 weeks prior to registration
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine < 2.0 mg/dL
* Bilirubin < 2 mg/dL (may be up to 3.0 mg/dL if due to liver involvement by lymphoma)

EXCLUSION CRITERIA:

* Prior chemotherapy or radiation therapy for lymphoma
* Prior anthracyclines or platinum compounds used as systemic chemotherapy
* Prior radiation therapy to the mediastinum or to ≥ 25% of the bone marrow
* Concurrent pentostatin or trastuzumab (Herceptin®)
* Pregnant or nursing
* Prior malignancy within the past 5 years unless it was in situ OR was treated with curative intent AND the patient has remained relapse-free
* HIV positive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (104):
- United States (104):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Horning SJ, Juweid ME, Schoder H, Wiseman G, McMillan A, Swinnen LJ, Advani R, Gascoyne R, Quon A. Interim positron emission tomography scans in diffuse large B-cell lymphoma: an independent expert nuclear medicine evaluation of the Eastern Cooperative Oncology Group E3404 study. Blood. 2010 Jan 28;115(4):775-7; quiz 918. doi: 10.1182/blood-2009-08-234351. Epub 2009 Sep 18. PMID 19767508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Eastern Cooperative Oncology Group (ECOG) member institutions between 4/7/2006 and 8/5/2009. The first patient was accrued on 9/26/2006.
Groups:
- Group I (PET Positive): Initially, patients received Rituximab 375 mg/m2 IV Day 1, Cyclophosphamide 750 mg/m2 IV Day 1, Vincristine 1.4 mg/m2 (max: 2 mg) IV Day 1, Doxorubicin 50 mg/m2 IV Day 1, and Prednisone 100 mg/m2 PO Days 1-5 (R-CHOP) every 21 days for 4 cycles. PET scan and conventional restaging occurred between days 14-20 of cycle 3. Patients who were PET positive after 3 cycles of R-CHOP received Rituximab 375 mg/m2 IV Day 1, Ifosfamide 5000 mg/m2 IV over 24 hours Day 2, Carboplatin AUC 5 (max: 800 mg) IV Day 2, Etoposide 100 mg/m2 IV Days 1, 2, 3 (R-ICE), Mesna 5000 mg/m2 IV over 24 hours Day 2, and Filgrastim 5 mcg/kg/day subcutaneous (SC) Day 4 until absolute neutrophil count (ANC) recovery every 14 days for 4 cycles .
- Group II (PET Negative): Initially, patients received Rituximab 375 mg/m2 IV Day 1, Cyclophosphamide 750 mg/m2 IV Day 1, Vincristine 1.4 mg/m2 (max: 2 mg) IV Day 1, Doxorubicin 50 mg/m2 IV Day 1, and Prednisone 100 mg/m2 PO Days 1-5 (R-CHOP) every 21 days for 4 cycles. PET scan and conventional restaging occurred between days 14-20 of cycle 3. Patients who were PET negative after 3 cycles of R-CHOP received 2 more cycles of R-CHOP (6 cycles in total).
- No Mid-Treatment PET: Initially, patients received Rituximab 375 mg/m2 IV Day 1, Cyclophosphamide 750 mg/m2 IV Day 1, Vincristine 1.4 mg/m2 (max: 2 mg) IV Day 1, Doxorubicin 50 mg/m2 IV Day 1, and Prednisone 100 mg/m2 PO Days 1-5 (R-CHOP) every 21 days for 4 cycles. PET scan and conventional restaging occurred between days 14-20 of cycle 3. Patients who did not have mid-treatment PET scan for any reasons came off study and continued to be followed up for disease progression and survival.
Period: Step 1 (R-CHOP X 3 Cycles)
Arm/Group | Group I (PET Positive) | Group II (PET Negative) | No Mid-Treatment PET
Started | 17 | 77 | 6
Treated | 17 | 77 | 5
Eligible and Treated | 13 | 63 | 4
Completed | 13 | 63 | 0
Not Completed | 4 | 14 | 6
Not completed — Patient ineligible | 4 | 14 | 1
Not completed — Did not start treatment | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other complicating disease | 0 | 0 | 1
Period: Step 2 (Tx Based on Mid-treatment PET)
Arm/Group | Group I (PET Positive) | Group II (PET Negative) | No Mid-Treatment PET
Started | 17 (All patients who started step 2 therapy were included regardless of eligibility.) | 76 (One patient withdrew from the study after step 1 treatment.) | 0
Eligible and Treated | 13 | 61 | 0
Completed | 10 | 58 | 0
Not Completed | 7 | 18 | 0
Not completed — Patient ineligible | 4 | 15 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other complicating disease | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Alternative therapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (PET Positive) | Group II (PET Negative) | No Mid-Treatment PET | Total
Number analyzed (Participants) | 13 | 63 | 4 | 80
Age, Continuous [Median (Full Range); unit: years] | 61 [20 to 70] | 63 [36 to 74] | 54 [33 to 60] | 62 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 28 | 2 | 34
  Male | 9 | 35 | 2 | 46

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-Free Survival (PFS)
Description: 2-year progression-free survival is defined as the probability of patients who remain alive and progression free at 2 years from study entry. The method of Kaplan and Meier (1958) was used to estimate PFS.
Time Frame: Assessed every 4 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, then every 12 months if patient is 5-10 years from study entry.
Measure: Number (90% Confidence Interval); unit: probability
Groups:
- Group I (PET Negative): Eligible and treated patients who were PET negative after 3 cycles of R-CHOP received 2 more cycles of R-CHOP (6 cycles in total).
- Group II (PET Positive): Eligible and treated patients who were PET positive after 3 cycles of R-CHOP received 4 cycles of R-ICE.
Arm/Group | Group I (PET Negative) | Group II (PET Positive)
Number analyzed (Participants) | 61 | 13
probability | 0.76 [0.65 to 0.84] | 0.42 [0.19 to 0.63]

2. Secondary Outcome: 5-year Overall Survival
Description: 5-year overall survival is defined as the probability of patients who remain alive at 5 years from study entry. The method of Kaplan and Meier (1958) was used to estimate overall survival.
Time Frame: Every 4 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, then every 12 months if patient is 5-10 years from study entry.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Group I (PET Negative) | Group II (PET Positive)
Number analyzed (Participants) | 61 | 13
probability | 0.77 [0.49 to 0.91] | 0.69 [0.43 to 0.85]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on R-CHOP treatment and every 2 weeks while on R-ICE treatment, and for 30 days after the end of treatment, up to 24 weeks.
Groups:
- Step 1 - All Treated Patients: All treated patients regardless of eligibility.
- Step 2 - Mid-treatment PET Positive: Patients who were mid-treatment PET positive and who received R-ICE in step 2 regardless of eligibility.
- Step 2 - Mid-treatment PET Negative: Patients who were mid-treatment PET negative and who received additional R-CHOP in step 2 regardless of eligibility.
Arm/Group | Step 1 - All Treated Patients | Step 2 - Mid-treatment PET Positive | Step 2 - Mid-treatment PET Negative
Serious Adverse Events (participants affected / at risk) | 58/99 | 17/17 | 25/76
Other Adverse Events (participants affected / at risk) | 97/99 | 17/17 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - All Treated Patients (N=99) | Step 2 - Mid-treatment PET Positive (N=17) | Step 2 - Mid-treatment PET Negative (N=76)
Anemia (Blood and lymphatic system disorders) | 5 | 7 | 5
Leukocytes decreased (Investigations) | 35 | 10 | 14
Lymphopenia (Investigations) | 9 | 8 | 6
Neutrophils decreased (Investigations) | 41 | 11 | 12
Platelets decreased (Investigations) | 8 | 15 | 5
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Fatigue (General disorders) | 4 | 1 | 1
Fever w/o neutropenia (General disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Weight gain (Investigations) | 1 | 0 | 0
Coagulation-other (Investigations) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Perforation, small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 0 | 3
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 1 | 0
Infection w/ gr3-4 neut, peritoneal (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 1 | 0 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0 | 0
Infection w/ gr3-4 neut, vulva (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, joint (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, larynx (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 0 | 1 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Head/headache (Nervous system disorders) | 1 | 0 | 0
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - All Treated Patients (N=99) | Step 2 - Mid-treatment PET Positive (N=17) | Step 2 - Mid-treatment PET Negative (N=76)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 73 | 16 | 57
Leukocytes decreased (Investigations) | 39 | 8 | 25
Lymphopenia (Investigations) | 11 | 3 | 10
Neutrophils decreased (Investigations) | 25 | 3 | 8
Platelets decreased (Investigations) | 23 | 8 | 13
Hypertension (Vascular disorders) | 5 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Fatigue (General disorders) | 71 | 16 | 50
Fever w/o neutropenia (General disorders) | 0 | 4 | 2
Insomnia (Psychiatric disorders) | 27 | 2 | 6
Rigors/chills (General disorders) | 6 | 1 | 0
Weight loss (Investigations) | 6 | 0 | 0
Flushing (Vascular disorders) | 7 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 58 | 7 | 31
Injection site reaction (General disorders) | 0 | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 22 | 6 | 9
Constipation (Gastrointestinal disorders) | 52 | 3 | 14
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16 | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 6 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 9 | 3 | 4
Nausea (Gastrointestinal disorders) | 50 | 10 | 25
Salivary (Gastrointestinal disorders) | 0 | 1 | 0
Taste disturbance (Nervous system disorders) | 22 | 3 | 14
Vomiting (Gastrointestinal disorders) | 15 | 4 | 3
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 2 | 0
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 1 | 0
Edema limb (General disorders) | 5 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 1 | 8
Alkaline phosphatase increased (Investigations) | 22 | 7 | 4
Alanine aminotransferase increased (Investigations) | 12 | 3 | 9
Aspartate aminotransferase increased (Investigations) | 20 | 7 | 15
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 0 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 3 | 4
Creatinine increased (Investigations) | 5 | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 58 | 9 | 32
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 6 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic/Laboratory-other (Investigations) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 9 | 2 | 1
Extrapyramidal movement (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 50 | 6 | 39
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 9 | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Head/headache (Nervous system disorders) | 14 | 3 | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 14 | 0 | 0
Pain NOS (General disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 6
Fistula oral cavity (Gastrointestinal disorders) | 0 | 1 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Cystitis (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 5 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No